CLINICAL TRIAL: NCT06662487
Title: The Effect of Free Weight Resistance Training and Body Composition on Cognitive Function Explored Through Eye Tracking
Brief Title: The Effect of Free Weight Resistance Training and Body Composition on Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Valparaiso (Other)
Responsible Party: Principal Investigator, Carlos Cristi Montero, Head of Investigation, Pontificia Universidad Catolica de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BIOEPUCV-HB 546-2022
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Cognitive Performance
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Free Weight Resistance Training (FWRT) (Experimental): Participants in the experimental group will engage in a 10-week free weight resistance training program. This program will consist of 3 weekly sessions, including exercises such as squats, deadlifts, and bench presses, among others. The training will focus on progressively increasing the intensity, working within a range of 60% to 80% of the one-repetition maximum (1RM).
  Interventions: Behavioral: Resistance Training
- Control Group (No Intervention): Participants in the control group will not receive any intervention and will be instructed to continue with their usual daily routine. These participants will be evaluated pre- and post-intervention in the same manner as the experimental group but will not participate in the training program.

INTERVENTIONS:
Behavioral: Resistance Training — Participants in the experimental group will perform free weight resistance training sessions focused on push, pull, and leg movement patterns. The program will last for 10 weeks, progressively increasing in load and intensity. The intervention will be designed to improve the participants' physical strength and observe how these changes affect their cognitive performance.
  Arms: Free Weight Resistance Training (FWRT)

SUMMARY:
This study, titled The Effect of Free Weight Resistance Training (FWRT) on Cognitive Function Explored through Eye Tracking, will be a randomized double-blind clinical trial aimed at evaluating how FWRT influences cognitive processing in healthy young adults. Eye-tracking technology will be used to measure reading metrics and DXA scans will be used to measure body composition before and after a 10-week FWRT intervention.

Participants will be randomly assigned to either an experimental group, which will undergo a 10-week FWRT program, or a control group. This study will provide insights into the potential benefits of free weight resistance training on the cognitive performance of text processing tasks.

ELIGIBILITY:
Inclusion Criteria:

* University students between the ages of 18 and 30.
* Healthy individuals with no recent participation (last six months) in physical training programs.
* Normal or corrected-to-normal vision.

Exclusion Criteria:

* Physical or health limitations that prevent participation in a resistance training program.
* Current involvement in other physical training programs.
* Visual impairments that cannot be corrected with glasses or contact lenses.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Cognitive Measures (Eye-Tracking Metrics) | Up to 10 weeks post-intervention
  Cognitive metrics (as text processing metrics) will be measured through an eye-tracking device (EyeLink Portable Duo), with the following key metrics:
  * First Pass Reading Times: Total time spent on fixations during the first pass of reading within an area of interest.
  * Total Reading Times: The sum of the durations of all fixations within an area of interest, including revisits to previously read areas.
  * Other eye-tracking or comprehension measures could also be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Católica de Valparaíso,, Valparaíso, Chile